CLINICAL TRIAL: NCT05060523
Title: To Study Effect of the Combination of Midodrine and Tolvaptan Versus Tolvaptan Alone in Patients With Severe Hyponatremia in Cirrhosis(TOLMINA Trial) - An Open Label Placebo Randomized Control Trial
Brief Title: To Study Effect of the Combination of Midodrine and Tolvaptan Versus Tolvaptan Alone in Patients With Severe Hyponatremia in Cirrhosis(TOLMINA Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-42
Record Dates: First submitted 2021-08-19; First posted 2021-09-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-08

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Tolvaptan; Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tolvaptan with Midodrine (Experimental)
  Interventions: Drug: Tolvaptan Tablets; Drug: Midodrine Oral Tablet
- Tolvaptan with Placebo (Active Comparator)
  Interventions: Drug: Tolvaptan Tablets; Other: Placebo

INTERVENTIONS:
Drug: Tolvaptan Tablets — • Tolvaptan15 mg once a day for 7 days, stat with 7.5 mg and titrate to 15 mg in 24 hours max30 mg
Drug: Midodrine Oral Tablet — • Midodrine 5 mg at "0" hours and then 5 mg every 8 hours to maintain Target MAP-80
  Arms: Tolvaptan with Midodrine
Other: Placebo — Placebo of Midodrine
  Arms: Tolvaptan with Placebo

SUMMARY:
In this randomized controlled trial , The patients who satisfy the below inclusion and exclusion criteria will be included and they will be randomised, according to 2 groups ( in total 110patients in each group) to receive either Midodrine+Tolvaptan or tolvaptan+placebo for 7 days followed by follow up for 1 month. These patients will be admitted to the hospital from OPD or emergency.

In patients with cirrhosis with Patients with cirrhosis -there are two types of hyponatremia. hyponatremia is due to important losses of extracellular fluid, most commonly from the kidneys (because of overdiuresis due to treatment with excessive doses of diuretics) or from the gastrointestinal tract( hypovolemic hyponatremia) hyponatremia develops in the setting of expanded extracellular fluid volume and plasma volume with ascites and edema.This condition is known as hypervolemic or dilutional hyponatremia.A marked impairment of renal solute-free water excretion, resulting in disproportionate renal retention of water with respect to sodium retention.In SALT trail showed that tolvaptan showed improvement in Na+ concentration from baseline at 4 ,30 day. It acts on by increasing free water generation by blocking ADH receptors in distal convoluted tubule. A study by Patel et al in 2017 showed that midodrine also increasing the Na+ by increasing the free water delivery to distal convoluted tubules(in cirrhosis usually there is less water delivery to distal convoluted tubules in view of less GFR).Till now there is no study has been done as combination of midodrine and tolvaptan whether superior to tolvaptan alone or not .So our aim is to study combination of midodrine and tolvaptan verses tolvaptan alone in patients with hyponatremia.

DETAILED DESCRIPTION:
1. Aim and Objective -

   AIM:

   • To study effect of the combination of Midodrine and Tolvaptan versus Tolvaptan alone in patients with severe hyponatremia in cirrhosis.

   PRIMARY Objective :

   • To study the Improvement in sodium concentration from base line to target level 125 meq/L in patients with hyponatremia ( Time frame-1 week) SECONDARY Objective :- To study the

   1 The change in Na+ concentration at D2,D4,D5. 2) Maintenance of Na concentration at d14, d30 3) Improvement in Na+ concentration from base line to 130 meq/l at day 7 4) Improvement in ascites at day 7,30 5) Development of AKI, HE [ 1 week,2 weeks,D30] 6) Osmolality changes, urine volume,urinay Na + excretion at D3,D5,D7,D14 D30 7) Mean arterial pressure at D1,D7,D14,D30. 8) RBC water and Na concentration in RBC cell at day 7, 30 9) Change in body weight at day 7, 30 10) The urine metabolomics
2. Methodology:

   * Study Definitions:

Hyponatermia as

Mild-126-130 Moderate-121-125 Severe-<120 Acute-<48 hours Chronic >48 hours - alukal et al 2020 Symptomatic-presence of symptoms Asymptomatic-no symptoms

Study population -All the patients of cirrhosis of liver patients visiting to ILBS and diagnosed to have hyponatremia Study design - Open label Placebo RCT

Assuming that the response rate is 30% in tolvaptan group and 50% in midodrine +tolvaptan group Alpha Error-5%,power 80% we need to enroll 200 cases, 100 each group.Further assuming 10% drop rate, 220 cases-110 in each arm(Allocated each group block randomization method, block size-10)

At baseline, a complete history with clinical and physical examination, a record of demographic profile, standard of care biochemical investigations would be done. All included patients will be evaluated with -

* Etiology of cirrhosis
* Upper GI endoscopy
* Haemogram (including reticulocyte count)
* Liver function tests,Renal function tests
* CBC/LFT/KFT/ELECTOLYTES/URINENa,URINEOsmolality,Sosmolality,thyroidprofile,S Cortisol,S ADH,RBC water,RBC Na
* UGIE endoscopy,Usg Abdomen/IVC and 2D echo,cardichaemodynamics,PRO BNP,PRA, Renal resistivity index
* USG abdomen with Doppler study
* Fibroscan
* Child-Pugh score , MELD The patients will be managed according to randomization. Subsequently, patients would be assessed clinically each day at the baseline and post-treatment at every day for 1 month.

ADVERSE EFFECTS Thirst Dry mouth Hypernatremia Renal dysfunction Abdomnal pain Nasea/Vomitting Muscle cramp

DURATION:

ELIGIBILITY:
Inclusion Criteria:

1. Child B/C cirrhosis
2. Hyponatremia( severe)
3. Written informed consent
4. Age-18-70 years

Exclusion Criteria:

1. AKI(1.5mg/dl)
2. Sepsis
3. Underlyig CKD
4. High risk varices
5. Recent Bleed in 2 weeks
6. Acute Symptomatic hyponatremia
7. SIADH
8. Hypothyroidism
9. Severe cardiopulmonary disease
10. Cerebrovascular accident
11. Multiple strokes;
12. Pseudohyponatremia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-09-19 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in Na+ to 125meq/L | 1 week

SECONDARY OUTCOMES:
Improvement in Na + (120 -125 meq/L) | 3 days
Improvement in Na + (120 -125 meq/L) | 5 days
Changes in Serum osmolality | 0,1day,3day,1week ,2 week,1 month
  Serum osmolality normal range is 285 to 295 millimol/kg
Changes in urine volume | 0,1day,3day,1week ,2 week,1 month
Changes in urinay Na + excretion in body | 0,1day,3day,1week ,2 week,1 month
Change in clinical complications(AKI,HE) in patients with hyponatremia | 1 week,1month
Development of AKI | 7 day
  Changes is serum creatine level more than 0.3 within 24 hours
Failure to achieve sodium concentration to 125 meq/L | 7 day
Improvement in Na+ concentration from base line to 130 meq/l | Day 7
Mean Arterial pressure | Day 1,7,14, and 30
sodium concentration in RBC cell | Day 7
  It is measured by calorimetry
sodium concentration in RBC cell | Day 30
  It is measured by calorimetry
RBC water concentration in RBC cell | Day 7
  It is measured by calorimetry
RBC water concentration in RBC cell | Day 30
  It is measured by calorimetry
Improvement in ascites | Day 30
  I t will be measured by ultrasound abdomen and graded as Grade 1 (Mild) , Grade 2 (moderate) & Grade 3 (massisve)
Maintenance of sodium concentration | Day 14 and 30
Change in body weight | Day 7
  It is measured by kilograms
Change in body weight | Day 30
  It is measured by kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided